CLINICAL TRIAL: NCT06689553
Title: A Multi-Center, Multinational, Prospective, Open-Label, Single Arm, Pilot Study to Assess the Feasibility, Safety and Tolerability of a Percutaneously Delivered Automated Continual Fluid Removal System in Patients With Advanced Diuretic-Resistant Heart Failure
Brief Title: Percutaneously Delivered Automated Continual Fluid Removal System in Patients With Advanced Diuretic-Resistant Heart Failure
Acronym: CLEAR-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paragate Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM10002
Record Dates: First submitted 2024-11-05; First posted 2024-11-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal implanted device (Experimental): Implantation and activation of an automated continual water removal system
  Interventions: Device: Automated Continual Fluid Removal System

INTERVENTIONS:
Device: Automated Continual Fluid Removal System — The intraperitoneal device is percutaneously implanted via mini laparotomy, under local anaesthesia and sedation, and connected to the wearable rechargeable pump through extracorporeal tubing. The device aims to remove excess fluids in heart failure patients with diuretic resistance

SUMMARY:
The study aims to assess the feasibility, safety, tolerability and functionality of a percutaneously delivered automated continual fluid removal System in up to 8 patients with Heart Failure (HF) and diuretic resistance.

Intervention: Implanted absorption chamber, connected to an external pump. Follow up: 6 months post activation.

DETAILED DESCRIPTION:
Objectives: To assess the feasibility, safety, tolerability and functionality of an intra-peritoneal, mechanically induced ultrafiltration system (IPUDx), through the analysis of procedure and device related serious adverse events and device function.

Study Duration: Up to 24 months. Enrolment 15 months, Activation following implantation (per patient) up to 1 month, Follow-up (per patient) 6 months, Close-out 2 months.

Number of Subjects: Up to 8 Diagnosis and Main Inclusion Criteria: Patients with fluid overloaded congested heart failure (The New York Heart Association Class II-IV) with diuretic resistance and a history of multiple heart failure related admissions.

Study Centers: Up to 5 Medical Centers in Serbia and Spain.

Study Product and Planned Use: The Paragate Medical IPUDx System comprises an intraperitoneally implanted fluid absorption chamber with an external wearable rechargeable pump, drainage bag and controller.

The system induces isotonic fluid loss across the peritoneal membranes which is collected in the fluid absorption chamber and transported to a daily disposable external fluid drainage bag.

Statistical Methodology: No statistical hypothesis is proposed. Safety will be evaluated using a complete description of Serious Adverse Events (SAEs). A descriptive analysis will be performed for all primary and secondary variables of the study for the basal measures and all post-basal measures. Interim analysis for all the study endpoints will be performed at the completion of the active follow up phase (3 months post activation). Safety analysis for Adverse Device Effects (ADEs) will be performed both at 3-month post activation and at the completion of maintenance phase (6 months post implantation).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Life expectancy > 6 months
* Heart Failure, New York Heart Association (NYHA) class II-IV
* > 1 HF related admissions in the last 12 months
* Fluid congestion (2 signs of pitting oedema, jugular distention, BW elevation, nocturnal dyspnoea score, respiration rate, pulmonary congestion and/or pleural effusion per chest x-ray, ascites)
* Failure to achieve effective diuresis and congestion relief despite appropriate or escalating diuretic doses or combination of diuretics
* Able to give written informed consent
* Ability to comply with study procedures and ability to operate the device themselves or by a regular caregiver support
* Residence in proximity to the medical center to ensure easy access for required hospital visits and to enable home visits
* Women of childbearing potential should use adequate contraception for as long as the device is implanted

Exclusion Criteria:

* Any non-cardiac disease with life expectancy < 1 year
* Any patient listed for solid organ transplantation
* Patients with a history, or with an indication for mechanical circulatory support
* intravenous (IV) inotropes required in last 3 months (INTERMACS Score

  * 3), excluding Levosimendan
* Immunocompromised (e.g. chronic steroid treatment, Human immunodeficiency virus (HIV), etc.)
* Insulin dependent diabetes with evidence of infection
* Severe hyponatremia as defined by a serum Sodium < 120 mmol/l
* Serum Albumin < 2.5 g/Dl
* Glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 by MDRD method, using MDRD 4-variable equation that includes age, sex, ethnicity, and serum creatinine
* Previous significant intraabdominal surgery, severe abdominal adhesions, intra-abdominal foreign body (except for small inguinal mesh)
* Current or historical (within last 6 months) large diaphragmatic hernia, or surgically irreparable, complex or recurring hernia
* 6 minutes walk test of less than 100 meters in all repeated testing (if applicable), or similar test
* Severe, multiple repeated cardiac-related ascites, subject to principal investigator (PI) discretion
* Inflammatory or ischemic bowel disease (i.e., Crohn's disease, ulcerative colitis) and frequent episodes of diverticulitis
* Current gastrointestinal active infection in the body (such as Clostridium difficile infection)
* Gastrointestinal haemorrhage within the last 4 months
* Bacterial peritonitis episode within the last 24 months
* > 2 systemic or local infections, such as urinary tract infection or abdominal skin infection within the last 6 months
* Class B or C liver cirrhosis of non-cardiac aetiology
* 18.5 > body mass index (BMI) > 40 presenting a risk for surgery
* Patients with contraindications for general/local anaesthesia, sedation and

  * or Percutaneous / Laparoscopic surgery
* Unsuitability for self-maintenance of the experimental home set-up
* Presence of any current cancer, subject to PI discretion
* Presence of any active implantable or body-worn devices that cannot be removed excluding Implantable Cardioverter-Defibrillator (ICD) / pacemaker, subject to PI discretion
* Known hypersensitivity to Nitinol nickel/titanium alloy and brilliant blue
* Pregnancy
* Patients being in another therapeutic clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of AEs related to implantation | 3 months post activation
  based on analysis of the incidence of serious adverse events related to the implantation procedure.
Serious Adverse Events related to the device | 3 months post activation and 6 months from implantation
  Based on the incidence of serious adverse events related to the device
Successful Implantation Rate | 3 months post activation
  based on post-insertion imaging confirmation utilizing imaging modalities such as X-rays to confirm the appropriate placement and positioning of the chamber within the peritoneal cavity (appropriate placement yes/no)

SECONDARY OUTCOMES:
Device Functionality | 3 months post activation
  assessed by: Weekly measurements of fluid removal volume (ml)
Clinical assessment of fluid overload | 3 months post activation
  A composite score evaluating fluid overload, incorporating physical examination findings (e.g., presence of edema, jugular venous distension) and patient-reported symptoms. Each clinical sign will be assessed individually and aggregated into a composite score to quantify the degree of fluid overload, allowing assessment of the intervention's effectiveness in managing fluid balance over time
Effectiveness of the drainage fluid | 3 months post activation
  assessed by comparing the sodium concentration in the drained fluid to the sodium concentration in the 24-hour urine collection and multiplying this ratio by the volume of the drained fluid
Echocardiographic assessment | 3 months post activation
  Evaluation of cardiac structure and function through echocardiographic imaging, with measurements including ventricular volumes, ejection fraction, and wall motion. These assessments will be aggregated to provide a comprehensive echocardiographic profile as a single outcome, focusing on overall cardiac function and structural changes over time
Quality of life questionnaire (KCCQ-12 questionnaire) | 3 months post activation
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period.
  KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
6 minutes' walk test | 3 months post activation
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Number of HF congestion related hospital admissions | 3 months post activation
  Tracking the frequency of hospital admissions specifically related to heart failure (HF) congestion, as an indicator of the device's impact on patient symptoms and management of HF-related complications
Dyspnoea Score | 3 months post activation
  assessed by using the Modified Borg Dyspnoea scale at rest - before and during 6 minutes walk test. This is a scale that asks the patient to rate the difficulty of his breathing. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal.
Markers of heart failure Severity: | 3 months post activation
  Measurement of specific biomarkers associated with heart failure severity, including NT-proBNP, Antigen carbohydrate 125, Cystatin C, and Interleukin-6, to assess the physiological impact of the intervention on HF progression and patient health status
Levels of Serum Creatinine | 3 months post activation
  Measurement of serum creatinine levels to evaluate kidney function and monitor potential changes associated with the intervention, providing insight into renal health in heart failure patients
Electrolytes levels | 3 months post activation
  Assessment of serum electrolyte levels (e.g., sodium, potassium), reported as a combined outcome with consistent units (e.g., mEq/L) to evaluate changes in electrolyte balance, which can reflect kidney function and fluid status in heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Marko Banović, MD, Principal Investigator — University Clinical Centre of Serbia; Marija Zdravkovic, MD, Principal Investigator — University Clinical Hospital Medical Center "Bezanijska kosa"
Locations (3):
- Serbia (2):
  - University Clinical Centre of Serbia, Belgrade, Visegradska 26
  - University Clinical Hospital Medical Center "Bezanijska kosa", Belgrade
- Hospital Clínico Universitario de Valencia-España, Valencia, Spain, Spain